CLINICAL TRIAL: NCT07046130
Title: Effect of Reducing Resistance Training Volume on the inter-and Intra-individual Response of Neuromuscular Parameters in Older Adults
Brief Title: Reduction in Resistance Training Volume and Neuromuscular Adaptations in Older Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Santos Lopes da Silva, PhD Student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VRSETS6070
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Sarcopenia in Elderly; Dynapenia
Keywords: Sarcopenia; Strength exercise; Muscle health
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Volume - 2 Sets and 1 Set (RV2SETS/RV1SET) (Experimental): This group will follow a reduced-volume training protocol in both legs, allowing for an intra-subject comparison. One leg will perform two sets per exercise (RV2SETS), and the other leg will perform only one set per exercise (RV1SET). This design will help assess whether neuromuscular adaptations can be maintained with lower training volume in older adults.
  These participants will train twice per week for 10 weeks, performing unilateral leg press and unilateral knee extension exercises with two different set volumes (1 vs. 2 sets), one for each leg.
  Interventions: Behavioral: Resistance Training
- Maintained Volume - 3 Sets (MV3SETS) (Active Comparator): This group will continue training with the same volume used during the initial phase of the study, which is three sets per exercise for both legs. This protocol aligns with standard resistance training guidelines for older adults aiming to promote strength and muscle maintenance.
  These participants will perform three sets of unilateral leg press and unilateral knee extension exercises, twice per week, for 10 weeks.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — The mininum resistance training volume (12 sets/week) will be applied.

SUMMARY:
The goal of this clinical trial is to evaluate how reducing resistance training volume affects neuromuscular adaptations in older adults aged 60 to 70 years. The main questions it aims to answer are:

Can strength and muscle adaptations be maintained with lower training volume?

Does reducing training volume influence muscle power and hypertrophy in older adults?

Researchers will compare two groups:

A group that reduces training volume in one or both legs

A group that maintains the same training volume in both legs to see if reducing volume leads to different neuromuscular outcomes.

Participants will:

Complete an initial 10-week strength training program (2x/week) using unilateral leg press and knee extension machines, performing 3 sets per exercise

Undergo tests for muscle strength (1-RM), muscle thickness (ultrasound), and power (isokinetic dynamometry) at weeks 0, 5, and 10

After 10 weeks, be randomly assigned to:

A reduced-volume group: one leg does 2 sets and the other 1 set per exercise

Or a control group: both legs continue doing 3 sets

Continue training for another 10 weeks under the assigned protocol

Repeat strength, muscle thickness, and power assessments at weeks 5 and 10 of phase 2

Attend a dietary intake interview with a registered dietitian

This study will help determine the minimum effective training volume needed to maintain strength and muscle health in older adults, potentially improving long-term adherence to exercise programs.

DETAILED DESCRIPTION:
Aging is associated with a progressive decline in muscle strength, muscle mass, and power, which can negatively affect functional capacity and quality of life in older adults. Resistance training (RT) is widely recognized as an effective intervention to mitigate these neuromuscular declines; however, adherence and long-term sustainability of high-volume RT programs can be challenging in this population due to reduced recovery capacity and potential lifestyle constraints. In this context, identifying the minimum effective training volume necessary to maintain neuromuscular adaptations is essential, as lower volumes may increase adherence among older adults. Therefore, this randomized, controlled clinical trial aims to investigate the effect of reducing RT volume on neuromuscular outcomes in older adults aged 60 to 70 years. The study will be conducted in two phases. In Phase 1, all participants will complete a 10-week RT program (2 sessions/week), performing three sets of unilateral leg press and knee extension exercises, with assessments of strength (1RM), muscle thickness (via ultrasound), power (via isokinetic dynamometry), body composition (via DXA), and dietary intake (via 24-hour recall) conducted at baseline, week 5, and week 10. Participants will be familiarized with the training procedures, and reliability in strength testing will be confirmed prior to the intervention. In Phase 2, participants will be randomized according to the delta (%) change in knee extension 1RM and assigned to one of two groups: a reduced-volume group, in which one leg performs two sets and the other one set (intra-subject design), or a control group maintaining three sets per leg. This second phase will also last 10 weeks, with follow-up assessments at weeks 5 and 10. The unilateral training design allows for within-subject comparisons to assess the impact of reduced volume, and the control group allows for between-group analysis, facilitating the identification of individual responses and determining whether neuromuscular adaptations can be maintained with lower training volumes after a standard RT protocol.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 60 and 70 years
* No participation in a regular resistance training program in the past six months
* Cleared for physical activity according to the Physical Activity Readiness Questionnaire (PAR-Q)

Exclusion Criteria:

* Musculoskeletal limitations that prevent participation in the training program
* Uncontrolled systemic arterial hypertension (resting systolic blood pressure >160 mmHg and/or diastolic >90 mmHg)
* Uncontrolled chronic diseases (e.g., heart failure, kidney disease, type 2 diabetes mellitus)
* Current diagnosis of cancer
* Unintentional weight loss of more than 3 kg in the past three months

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-12-18 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Maximum Dynamic Strength (1-RM) in Knee Extension and Leg Press (kg) | Up to end of study data collection (both stages), i.e., assessed up to 1 year
  This measurement will be assessed in both stages of the study.
  In Phase 1 (initial training), 1-RM testing will be performed for unilateral knee extension and unilateral leg press exercises. After a familiarization session, participants will complete up to three testing sessions, 72 hours apart, until consistent values (≤5% variation) are reached. Assessments will be conducted at baseline (week 0), mid-intervention (week 5), and post-intervention (week 10).
  In Phase 2 (volume manipulation), 1-RM measurements will be repeated at weeks 5 and 10, following the same standardized testing procedures. All evaluations will be performed at least 72 hours after the last training session to minimize the influence of acute fatigue on strength performance.

SECONDARY OUTCOMES:
Muscle Thickness (cm) - Quadriceps Muscle Group (Ultrasound) | Up to end of study data collection (both stages), i.e., assessed up to 1 year
  This measurement will be assessed in both stages of the study.
  In Phase 1, muscle thickness of the quadriceps will be measured by B-mode ultrasound imaging at baseline (week 0), mid-intervention (week 5), and post-intervention (week 10). Measurements will be performed on both legs following a standardized protocol, with the participant in a rested state.
  In Phase 2, the same procedure will be followed to reassess muscle thickness at weeks 5 and 10, with all evaluations occurring at least 72 hours after the last training session to reduce the influence of acute changes in muscle size.
Thigh Fat-Free Mass (kg) - Dual-Energy X-ray Absorptiometry (DXA) | Up to end of study data collection (both stages), i.e., assessed up to 1 year
  This measurement will be assessed in both stages of the study.
  Thigh fat-free mass will be evaluated by DXA scan at five time points: baseline (week 0), mid-intervention (week 5), and post-intervention (week 10) of Phase 1, as well as at week 5 and week 10 of Phase 2. Scans will be performed using a standardized protocol by trained technicians. Participants will be instructed to avoid vigorous physical activity and follow pre-assessment guidelines for 24 hours prior to each scan to ensure consistent and reliable measurements.
Average Power (Watts) - Isokinetic Knee Extension Test | Up to end of study data collection (both stages), i.e., assessed up to 1 year
  This measurement will be assessed in both stages of the study.
  Power of the knee extensors will be measured using an isokinetic dynamometer during concentric unilateral knee extension at standardized angular velocities. Assessments will be performed at baseline (week 0), mid-intervention (week 5), and post-intervention (week 10) in both phases.
  All power assessments will be conducted at least 72 hours after the last training session to minimize the effects of fatigue and ensure valid measures of peak performance.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education and Sports of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No